CLINICAL TRIAL: NCT00933270
Title: Comparison of the SUpera® PERipheral System to a Performance Goal Derived From Balloon Angioplasty Clinical Trials in the Superficial Femoral Artery
Brief Title: Comparison of the SUpera® PERipheral System in the Superficial Femoral Artery
Acronym: SUPERB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Baim Institute for Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SFA-1 US/EU
Record Dates: First submitted 2009-07-02; First posted 2009-07-07 (Estimated); Results first posted 2015-03-25 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Peripheral Vascular Disease
Keywords: Superficial Femoral Artery or SFA
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SUPERA® Nitinol Stent System (Experimental): Implantation of SUPERA nitinol stent using the SUPERA® Nitinol Stent System
  Interventions: Device: SUPERA® Nitinol Stent System

INTERVENTIONS:
Device: SUPERA® Nitinol Stent System — Percutaneous Angioplasty of the Superior Femoral Artery with placement of a SUPERA® Stent at time of PTA

SUMMARY:
This is a prospective, multicenter, non-randomized, single arm, pivotal trial.

The main objective of this study is to demonstrate the safety and effectiveness of the IDev SUPERA® Nitinol Stent System in treating subjects with obstructive superficial femoral artery (SFA) disease. The primary endpoint will be the primary patency of the SFA evaluated at 12 months. The outcome will be compared to a performance goal based on clinical trials of percutaneous transvenous angioplasty (PTA) alone.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years and of age of legal consent.
2. Women of child bearing potential must have a negative pregnancy test within 7 days prior to the index procedure.
3. Subject has lifestyle limiting claudication or rest pain (Rutherford-Becker scale 2-4) with a resting ankle-brachial index (ABI) less than or equal to 0.9. TBI (toe-brachial index) is performed only unable to assess ABI. TBI must be less than or equal to 0.7.
4. A single superficial femoral artery lesion with greater than 60% stenosis or total occlusion.
5. Stenotic lesion(s) or occluded length within the same vessel (one long or multiple serial lesions) greater than or equal to 40 mm to less than or equal to 140 mm. Reference vessel diameter (RVD) greater than or equal to 4.0 mm and less than or equal to 6.0 mm by visual assessment.
6. All lesions are to be located with the distal point at least 3 cm above the knee joint, defined as the distal end of the femur at the knee joint, and proximal point at least 2 cm below the origin of the profunda artery.
7. Patent infrapopliteal and popliteal artery, i.e., single vessel runoff or better with at least one of three vessels patent (less than 50% stenosis) to the ankle or foot.
8. The target lesion(s) can be successfully crossed with a guide wire and dilated.
9. Poor aortoiliac or common femoral "inflow" (i.e., angiographically defined greater than 50% stenosis of the iliac or common femoral artery) that would be deemed inadequate to support a femoropopliteal bypass graft must be successfully treated prior to treatment of the target lesion. This can be done just prior to treatment of the target lesion. Successful treatment is defined as less than 30% stenosis after either PTA or stenting of the inflow lesion. After treatment of the inflow lesion, the pressure gradient across the target lesion will be obtained and if the pressure gradient is greater than or equal to 20 mmHg, then the subject will be included in the study.
10. A subject with bilateral obstructive SFA disease is eligible for enrollment into the study. If a subject with bilateral disease is enrolled, the target limb will be selected at the Investigator's discretion, who may use the criteria of lesion length, percent stenosis, and/or calcification content. The contra-lateral procedure should not be done until at least 30 days after the index procedure (staged); however, if contralateral treatment is performed prior to treatment of the target lesion, the waiting period will be at least 14 days prior to the index procedure.
11. The subject is eligible for standard surgical repair, if necessary.
12. A subject who requires a coronary intervention should have it performed at least 7 days prior to the treatment of the target lesion.
13. Subject must provide written informed consent.
14. Subject must be willing to comply with the specified follow-up evaluation schedule.

Exclusion Criteria:

1. Thrombophlebitis or deep venous thrombus, within the previous 30 days.
2. Receiving dialysis or immunosuppressant therapy within the previous 30 days.
3. Thrombolysis of the target vessel within 72 hours prior to the index procedure, where complete resolution of the thrombus was not achieved.
4. Stroke within the previous 90 days.
5. Ipsilateral femoral aneurysm or aneurysm in the SFA or popliteal artery.
6. Required stent placement via a popliteal approach.
7. Required stent placement across or within 0.5 cm of the SFA/PFA bifurcation.
8. Procedures which are pre-determined to require stent-in-stent placement to obtain patency, such as in-stent restenosis.
9. Significant vessel tortuosity or other parameters prohibiting access to the lesion or 90° tortuosity which would prevent delivery of the stent device.
10. Required stent placement within 1 cm of a previously deployed stent.
11. Subject required a coronary intervention, and the coronary intervention was done less than 7 days prior to or planned within 30 days after the treatment of the target lesion.
12. Known allergies to any of the following: aspirin and all three of the following: clopidogrel bisulfate (Plavix®), ticlopidine (Ticlid®), and prasugrel (Effient®); heparin, nitinol (nickel titanium), or contrast agent, that cannot be medically managed.
13. Presence of thrombus prior to crossing the lesion.
14. Known or suspected active infection at the time of the procedure.
15. Presence of an ipsilateral arterial artificial graft.
16. Use of cryoplasty, laser, or atherectomy devices at the time of index procedure.
17. Restenotic lesion that had previously been treated by atherectomy, laser or cryoplasty within 3 months of the index procedure.
18. Subject has tissue loss, defined as Rutherford-Becker classification category 5 or 6.
19. History of neutropenia, coagulopathy, or thrombocytopenia that was unexplained or is considered to be at risk for reoccurrence.
20. Known bleeding or hypercoagulability disorder or significant anemia (Hb < 8.0) that cannot be corrected.
21. Subject has the following laboratory values:

    1. platelet count less than 80,000/μL,
    2. international normalized ratio (INR) greater than 1.5,
    3. serum creatinine level greater than 2.0 mg/dL.
22. Subject requires general anesthesia for the procedure.
23. Subject is pregnant or plans to become pregnant during the study.
24. Subject has a co-morbid illness that may result in a life expectancy of less than 1 year.
25. Subject is participating in an investigational study of a new drug, biologic or device at the time of study screening. NOTE: Subjects who are participating in the long term follow-up phase of a previously investigational and now FDA-approved product are not excluded by this criterion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2009-07; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol Base, RN,MS, Study Director — Abbott Medical Devices; Kenneth Rosenfield, MD, Principal Investigator — Massachusetts General Hospital; Lawrence Garcia, MD, Principal Investigator — Steward St. Elizabeth's Medical Center of Boston, Inc.
Locations (49):
- United States (49):
  - Cardiology Associates of Mobile, Inc., Fairhope, Alabama
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - Tucson Medical Center, Tucson, Arizona
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - ACT / CVRI & Cedar Sinai Medical Center, Beverly Hills, California
  - Hartford Hospital, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Bradenton Cardiology Center, Bradenton, Florida
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Mount Sinai Medical Cente, Miami Beach, Florida
  - Clarian North / Heart Partners, Fishers, Indiana
  - Cardiovascular Research of Northwest Indiana, LLC, Munster, Indiana
  - Hutchinson Hospital Corporation dba Promise Regional Medical Center, Hutchinson, Kansas
  - Willis Knighton Bossier Medical Center, Bossier City, Louisiana
  - Terrebonne General Hospital, Houma, Louisiana
  - Cardiovascular Institute of the South, Lafayette, Louisiana
  - Opelousas General Health System, Opelousas, Louisiana
  - Louisiana Heart Center, Slidell, Louisiana
  - Maine Medical Center, Portland, Maine
  - Montgomery General Hospital, Olney, Maryland
  - Massachussetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Caritas-St. Elizabeth Medical Center, Brighton, Massachusetts
  - Metro Health Hospital, Wyoming, Michigan
  - Hattiesburg Clinic, P.A., Hattiesburg, Mississippi
  - Deborah Heart, Browns Mills, New Jersey
  - Hunterdon Medical Center, Flemington, New Jersey
  - Robert Wood Johnson UMDNJ-RWJMS, New Brunswick, New Jersey
  - SJH Cardiology Associates, Liverpool, New York
  - NYU Medical Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - The Lindner Center for Research and Education at The Christ Hospital, Cincinnati, Ohio
  - University Hospital, Cleveland, Ohio
  - Ohio Health Research Institute / Riverside Methodist Hospital, Columbus, Ohio
  - Heritage Valley Health System, Beaver, Pennsylvania
  - Cardiology Consultants or Mainline Health System, Bryn Mawr, Pennsylvania
  - Moffitt Heart & Vascular Group, Wormleysburg, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - Greenville Hospital Systems, Greenville, South Carolina
  - Forsyth Medical Center - Cardiovascular Research, Winston-Salem, South Carolina
  - Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Vanderbilt Medical Center, Nashville, Tennessee
  - Alice Heart Center, Alice, Texas
  - Austin Heart, P.A, Austin, Texas
  - Cardiovascular Specialist of Texas & North Austin Medical Center, Austin, Texas
  - Cardiovascular Research Institute of Dallas, Dallas, Texas
  - Plaza Medical Center of Fort Worth, Fort Worth, Texas
  - North Cascade Cardiology, PLLC, Bellingham, Washington
  - Columbia - St. Mary's, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Palena LM, Isernia G, Parlani G, Veroux P, Ficarelli I, Frascheri A, Pischedda A, Patrone L, Dionisi CP, Cianni R, Airoldi F, Landino P, Kleiban A, Filauri P, Passalacqua G, Antignani PL, De Rose E, Valls A, Biondi-Zoccai G, Manzi M. A multicenter prospective observational study appraising the effectiveness of the Supera stent after subintimal recanalization of femoro-popliteal artery occlusion: The SUPERSUB II study. Catheter Cardiovasc Interv. 2024 May;103(6):963-971. doi: 10.1002/ccd.31028. Epub 2024 Apr 2. PMID 38566517
- [Derived] Garcia L, Jaff MR, Metzger C, Sedillo G, Pershad A, Zidar F, Patlola R, Wilkins RG, Espinoza A, Iskander A, Khammar GS, Khatib Y, Beasley R, Makam S, Kovach R, Kamat S, Leon LR Jr, Eaves WB, Popma JJ, Mauri L, Donohoe D, Base CC, Rosenfield K; SUPERB Trial Investigators. Wire-Interwoven Nitinol Stent Outcome in the Superficial Femoral and Proximal Popliteal Arteries: Twelve-Month Results of the SUPERB Trial. Circ Cardiovasc Interv. 2015 May;8(5):e000937. doi: 10.1161/CIRCINTERVENTIONS.113.000937. PMID 25969545

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 46 sites in the US enrolled 325 subjects into this study. The first patient was enrolled on July 30, 2009 and the last patient was enrolled on May 20, 2011. Intention-To-Treat (ITT) population included 264 subjects and Per-Protocol (PP) population included 257 subjects. In addition, 61 roll-in subjects were enrolled.
Groups:
- Supera® Peripheral Stent System: Implantation of Supera stent using the Supera® Peripheral Stent System
  Supera® Peripheral Stent System: Percutaneous Angioplasty of the Superficial Femoral or Proximal Popliteal Artery with placement of a Supera® Stent
Period: Overall Study
Arm/Group | Supera® Peripheral Stent System
Started | 264 (ITT population)
Completed | 177
Not Completed | 87
Not completed — Withdrawal by Subject | 26
Not completed — Insufficient Follow-up | 10
Not completed — Lost to Follow-up | 14
Not completed — Adverse Event | 1
Not completed — Missed Visit | 2
Not completed — Death | 24
Not completed — Moved or would not return | 10

BASELINE CHARACTERISTICS:
Population: The Intention-to-treat (ITT; n=264) analysis set included all subjects enrolled in the study excluding Roll-in subjects (n=61).
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 264
Age, Continuous [Mean (Standard Deviation); unit: years]
  ITT population | 68.7 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96
  Male | 168
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 244
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 35
  White | 221
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 264

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint: Freedom From Death, Target Lesion Revascularization (TLR), or Any Amputation of the Index Limb to 30 (±7) Days.
Time Frame: 30 days
Population: Per ITT set.
  Patients are included in the clinical endpoint if:
  * They return for their visit within the window
  * They came back for a later visit and the sponsor has information about their clinical status within the endpoint time frame
  * The last contact date predated the endpoint time frame but had an event within the endpoint time frame.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 260
percentage of participants
  Freedom from Death,TLR or amputation (30 days) | 99.2 [97.2 to 99.9]
  Freedom from All Cause Death to 30 days | 99.6 [97.9 to 100.0]
  Freedom from TLR to 30 days | 99.6 [97.9 to 100.0]
  Freedom from Amputation of the index limb(30 days) | 100.0 [98.6 to 100.0]

2. Primary Outcome: Primary Efficacy Endpoint: SFA Patency at 12 Months (± 30 Days), Defined as Freedom From Restenosis (PSVR ≥ 2.0) and TLR.
Description: Patency of the target lesion was defined as no evidence of restenosis or occlusion within the originally treated lesion based on a centrally-read Color Flow Doppler ultrasound in the absence of target lesion revascularization (TLR). Occlusion and restenosis were defined as no color flow or an increase in peak systolic velocity of > 2.0 when compared to the proximal normal segment.
Time Frame: 12 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 228
percentage of participants
  Patency rate at 12 months | 78.9 [73.1 to 84.1]
  No restenosis at 12 months | 86.7 [81.6 to 90.9]
  Freedom from TLR at 12 months | 88.9 [84.2 to 92.6]

3. Secondary Outcome: Technical (Lesion) Success
Description: Technical (lesion) success, defined as the attainment of <50% residual stenosis by Quantitative Angiography (QA) by any percutaneous method as determined by the Angiographic core laboratory.
Time Frame: intraoperative
Population: Per ITT set: Post-procedure angiogram analyzed by core lab
Measure: Number (95% Confidence Interval); unit: percentage of treated segments
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 262
percentage of treated segments | 100.0 [98.6 to 100.0]

4. Secondary Outcome: Procedural Success
Description: Defined as device success with < 50% residual stenosis immediately after stent placement, mean trans-stenotic pressure gradient less than 5 mmHg, and without the occurrence of death, amputation or repeat revascularization of the target lesion during the hospital stay.
Time Frame: intraoperative
Population: Per ITT set. Supera implanted. Post-procedure angiogram analyzed by core lab Occurrence of death, amputation or TLR during the hospital stay
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 261
percentage of participants | 100.0 [98.6 to 100.0]

5. Secondary Outcome: Device Success
Description: Device success, defined as achievement of a final residual diameter stenosis of <50% (by QA), using the assigned treatment only.
Time Frame: intraoperative
Population: Per ITT set: Supera implanted. Post-procedure angiogram analyzed by core lab
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 261
percentage of participants | 98.5 [96.1 to 99.6]

6. Secondary Outcome: Secondary Safety Composite Endpoint
Description: Secondary safety endpoint was a combined rate of death at 30 (± 7) days, or TLR, index limb amputation, and an increase in Rutherford-Becker Classification by 2 classes at 12 months (± 30 Days) (comparing pre- to post-procedural assessments).
Time Frame: 12 months (± 30 Days)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 233
percentage of participants | 12.45 [8.50 to 17.38]

7. Secondary Outcome: Secondary Safety Endpoint
Description: Secondary safety endpoint was a combined rate of death at 30 (± 7) days, or TLR, index limb amputation, and an increase in Rutherford-Becker Classification by 2 classes (comparing pre- to post-procedural assessments).
Time Frame: 24 months (± 30 Days)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 213
percentage of participants | 19.25 [14.18 to 25.19]

8. Secondary Outcome: Secondary Safety Endpoint
Description: Secondary safety endpoint was a combined rate of death at 30 (± 7) days, or TLR, index limb amputation, and an increase in Rutherford-Becker Classification by 2 classes at 36 months (± 30 Days)(comparing pre- to post-procedural assessments).
Time Frame: 36 months (± 30 Days)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 178
percentage of participants | 24.16 [18.07 to 31.13]

9. Secondary Outcome: Long-Term Safety Endpoint (Clinically Driven TLR, Index Limb Amputation)
Time Frame: 12 months (± 30 Days)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 235
percentage of participants | 11.5 [7.7 to 16.3]

10. Secondary Outcome: Long-Term Safety Endpoint (Clinically Driven TLR, Index Limb Amputation)
Time Frame: 24 months (± 30 Days)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 215
percentage of participants | 17.7 [12.8 to 23.4]

11. Secondary Outcome: Long-Term Safety Endpoint (Clinically Driven TLR, Index Limb Amputation)
Time Frame: 36 months (± 30 Days)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 184
percentage of participants | 22.3 [16.5 to 29.0]

12. Secondary Outcome: Stent Fracture Rate
Description: Stent fractures were analyzed by X-ray evaluation by a designated core laboratory and defined as type I, II, III, IV or V.
  Stent fracture classification
  * Type I - a single strut fracture only.
  * Type II - multiple single nitinol stent fractures that can occur at different sites.
  * Type III - multiple nitinol stent fractures resulting in complete transverse linear fracture but without stent displacement.
  * Type IV - a complete transverse linear type III fracture with stent displacement.
  * Type V - a spiral dissection of a stent.
Time Frame: 12 months (± 30 Days)
Population: Per ITT set: Supera implanted. Patient returned for visit and had x-ray of stent. X-ray analyzed by core lab
Measure: Number; unit: percentage of participants
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 244
percentage of participants
  Single Strut | 0
  Multiple Strut | 0
  Fragments Aligned | 0
  Fragments Malaligned | 0
  Spiral Fracture | 0

13. Secondary Outcome: Stent Fracture Rate
Description: Stent fractures were analyzed by X-ray evaluation by a designated core laboratory and defined as type I, II, III, IV or V.
Time Frame: 24 months (± 30 Days)
Population: Per ITT set: Supera implanted. Patient returned for visit and had x-ray of stent. X-ray analyzed by core lab
Measure: Number; unit: percentage of participants
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 202
percentage of participants
  Single Strut | 0
  Multiple Strut | 0
  Fragments Aligned | 0.5
  Fragments Malaligned | 0
  Spiral Fracture | 0

14. Secondary Outcome: Stent Fracture Rate
Description: as for outcome 13
Time Frame: 36 months (± 30 Days)
Population: Per ITT set: Supera implanted. Patient returned for visit and had x-ray of stent. X-ray analyzed by core lab
Measure: Number; unit: percentage of participants
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 162
percentage of participants
  Single Strut | 0
  Multiple Strut | 0
  Fragments Aligned | 0.6
  Fragments Malaligned | 0
  Spiral Fracture | 0

15. Secondary Outcome: Ankle-brachial Index (ABI) Measurements on Target Limb
Description: A ratio of the highest ankle systolic blood pressure in one leg, usually measured with a 10 cm cuff at the ankle and using a continuous wave Doppler to detect return of blood flow in the anterior tibial and posterior tibial arteries, to the highest of either arm systolic blood pressure. Performed at rest with subject in supine position.
Time Frame: Baseline
Population: Per ITT set: Baseline ABI measured prior to study procedure
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 257
ratio | 0.73 (0.18)

16. Secondary Outcome: Ankle-brachial Index (ABI) Measurements on Target Limb
Description: as for outcome 15
Time Frame: 1 month (± 7 Days)
Population: Per ITT set: Patient returned for visit and had ABI measured
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 251
ratio | 0.99 (0.17)

17. Secondary Outcome: Ankle-brachial Index (ABI) on Target Limb
Description: as for outcome 15
Time Frame: 6 Months (± 14 Days)
Population: Per ITT set: Patient returned for visit and had ABI measured
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 226
ratio | 0.92 (0.22)

18. Secondary Outcome: Ankle-brachial Index (ABI) on Target Limb
Description: as for outcome 15
Time Frame: 12 Months (± 30 Days)
Population: Per ITT set: Patient returned for visit and had ABI measured
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 227
ratio | 0.92 (0.22)

19. Secondary Outcome: Target Lesion Revascularization (TLR)
Description: Defined as any repeat percutaneous intervention with or without evidence of stenosis ≥ 50%, to improve blood flow inside or within 5 mm proximally and/or distally of the treated target lesion.
Time Frame: 6 months (± 14 Days)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 241
percentage of participants | 1.7 [0.5 to 4.2]

20. Secondary Outcome: Target Lesion Revascularization (TLR)
Description: as for outcome 19
Time Frame: 12 months (± 30 Days)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 235
percentage of participants | 11.1 [7.4 to 15.8]

21. Secondary Outcome: Target Lesion Revascularization (TLR)
Description: as for outcome 19
Time Frame: 24 months (± 30 Days)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 215
percentage of participants | 16.7 [12.0 to 22.4]

22. Secondary Outcome: Target Lesion Revascularization (TLR)
Description: as for outcome 19
Time Frame: 36 months (± 30 Days)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 183
percentage of participants | 21.3 [15.6 to 28.0]

23. Secondary Outcome: SFA Patency: PSV Ratio ≥ 2.0
Description: as for outcome 2
Time Frame: 6 Months (± 14 days)
Population: Per ITT set. Patients are included if: they return for visit within the window, returned for a later visit & sponsor has information on their clinical status within the endpoint time frame, the last contact date predated the endpoint time frame but had an event within the endpoint time frame, had a duplex ultrasound performed & analyzed by core lab
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 225
percentage of participants | 84.9 [79.5 to 89.3]

24. Secondary Outcome: SFA Patency: PSV Ratio > 2.4
Description: as for outcome 2
Time Frame: 6 Months (± 14 days)
Population: as for outcome 23
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 225
percentage of participants | 86.2 [81.0 to 90.4]

25. Secondary Outcome: SFA Patency: PSV Ratio > 2.4
Description: as for outcome 2
Time Frame: 12 Months (±30 days)
Population: Per ITT set. Patients are included if they return for visit within the window, returned for a later visit & sponsor has information on their clinical status within the endpoint time frame, the last contact date predated the endpoint time frame but had an event within the endpoint time frame, had a duplex ultrasound performed & analyzed by core lab
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 228
percentage of participants | 80.3 [74.5 to 85.2]

26. Secondary Outcome: Target Vessel Revascularization
Description: Defined as any repeat percutaneous intervention or bypass surgery performed in the target vessel at 6 months post-procedure.
Time Frame: 6 months (± 14 days)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 241
percentage of participants | 2.5 [0.9 to 5.3]

27. Secondary Outcome: Target Vessel Revascularization
Description: Defined as any repeat percutaneous intervention or bypass surgery performed in the target vessel at 12 months post-procedure.
Time Frame: 12 months (±30 days)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 235
percentage of participants | 13.2 [9.1 to 18.2]

28. Secondary Outcome: Target Vessel Revascularization
Description: Defined as any repeat percutaneous intervention or bypass surgery performed in the target vessel at 24 months post-procedure.
Time Frame: 24 months (±30 days)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 215
percentage of participants | 20.5 [15.3 to 26.5]

29. Secondary Outcome: Target Vessel Revascularization
Description: Defined as any repeat percutaneous intervention or bypass surgery performed in the target vessel at 36 months post-procedure.
Time Frame: 36 months (±30 days)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 186
percentage of participants | 25.8 [19.7 to 32.7]

30. Secondary Outcome: Limb Ischemia Improvement: Rutherford Becker Scale
Description: Defined as an improvement in the Rutherford-Becker Clinical Improvement Scale of greater than or equal to one.
  Grade +3 = Markedly improved. Symptoms are gone or markedly improved. ABI increased to >0.90.
  Grade +2 = Moderately improved. Still symptomatic but with improvement in lesion category. ABI increased by 0.10 but not normalized.
  Grade +1 = Minimally improved. Categorical improvement in symptoms without significant ABI increase (0.10 or less) or vice versa (but not both).
  Grade 0 = No change. No categorical shift and less than 0.10 change in ABI. Grade -1 = Mildly worse. Either worsening of symptoms or decrease in ABI of 0.10.
  Grade -2 = Moderate worsening. Deterioration of the subject's condition by one category or unexpected minor amputation.
  Grade -3 = Marked worsening. Deterioration of the subject's condition by more than one category or major amputation.
Time Frame: 1 month (± 7 days)
Population: Per ITT set.
  Patients are included in the Limb ischemia improvement if:
  They had a baseline Rutherford Becker Clinical Classification done. They return for their visit and Rutherford Becker Clinical Classification was done.
Measure: Number; unit: percentage of limbs
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 259
percentage of limbs | 97.3

31. Secondary Outcome: Limb Ischemia Improvement: Rutherford Becker Scale
Description: as for outcome 30
Time Frame: 12 Months (±30 days)
Population: as for outcome 30
Measure: Number; unit: percentage of limbs
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 230
percentage of limbs | 89.1

32. Secondary Outcome: Limb Ischemia Improvement: Rutherford Becker Scale
Description: as for outcome 30
Time Frame: 24 Months (±30 days)
Population: as for outcome 30
Measure: Number; unit: percentage of limbs
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 203
percentage of limbs | 89.2

33. Secondary Outcome: Limb Ischemia Improvement: Rutherford Becker Scale
Description: as for outcome 30
Time Frame: 36 Months (±30 days)
Population: as for outcome 30
Measure: Number; unit: percentage of limbs
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 167
percentage of limbs | 92.2

34. Secondary Outcome: Major Adverse Events (MAVE)
Description: Defined as a composite rate of
  1. stent thrombosis,
  2. clinically apparent distal embolization (defined as causing end-organ damage, e.g. lower extremity ulceration, tissue necrosis, or gangrene),
  3. procedure-related arterial rupture,
  4. acute limb ischemia,
  5. target limb amputation,
  6. procedure related bleeding event requiring transfusion.
Time Frame: 30 days (±7 days)
Population: Per ITT set. Patients are included if: they had a procedure related MAVE event, return for their visit within the window, returned for a later visit and the sponsor has information about their clinical status within the endpoint time frame, last contact date predated the endpoint time frame but had an event within the endpoint time frame.
Measure: Number; unit: percentage of participants
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 260
percentage of participants
  Stent Thrombosis | 0.4
  Clinically Apparent Distal Embolization | 0.4
  Procedure-Related Arterial Rupture | 0
  Acute Limb Ischemia | 0.4
  Target Limb Amputation | 0
  Procedure Related Bleeding Requiring Transfusion | 0.4

35. Secondary Outcome: Major Adverse Events (MAVE)
Description: as for outcome 34
Time Frame: 6 Months (±14 days)
Population: as for outcome 34
Measure: Number; unit: percentage of participants
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 241
percentage of participants
  Stent Thrombosis | 0.4
  Clinically Apparent Distal Embolization | 0.4
  Procedure-Related Arterial Rupture | 0
  Acute Limb Ischemia | 0.8
  Target Limb Amputation | 0
  Procedure Related Bleeding Requiring Transfusion | 1.2

36. Secondary Outcome: Major Adverse Events (MAVE)
Description: as for outcome 34
Time Frame: 12 months (±30 days)
Population: as for outcome 34
Measure: Number; unit: percentage of participants
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 235
percentage of participants
  Stent Thrombosis | 0.9
  Clinically Apparent Distal Embolization | 0.9
  Procedure-Related Arterial Rupture | 0
  Acute Limb Ischemia | 1.7
  Target Limb Amputation | 0.4
  Procedure Related Bleeding Requiring Transfusion | 1.3

37. Secondary Outcome: Major Adverse Events (MAVE)
Description: as for outcome 34
Time Frame: 24 months (±30 days)
Population: as for outcome 34
Measure: Number; unit: percentage of participants
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 209
percentage of participants
  Stent Thrombosis | 1.4
  Clinically Apparent Distal Embolization | 1.0
  Procedure-Related Arterial Rupture | 0
  Acute Limb Ischemia | 1.9
  Target Limb Amputation | 1.0
  Procedure Related Bleeding Requiring Transfusion | 1.4

38. Secondary Outcome: Major Adverse Events (MAVE)
Description: as for outcome 34
Time Frame: 36 months (±30 days)
Population: as for outcome 34
Measure: Number; unit: percentage of participants
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 175
percentage of participants
  Stent Thrombosis | 1.7
  Clinically Apparent Distal Embolization | 1.1
  Procedure-Related Arterial Rupture | 0
  Acute Limb Ischemia | 2.3
  Target Limb Amputation | 1.1
  Procedure Related Bleeding Requiring Transfusion | 1.7

39. Secondary Outcome: Index Limb Amputations
Description: Amputation was defined as the surgical removal of tissue anywhere from the toe to hip in the ipsilateral limb of the target site.
Time Frame: 6 months (±14 days)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 240
percentage of participants | 0 [0.0 to 1.5]

40. Secondary Outcome: Index Limb Amputations
Description: as for outcome 39
Time Frame: 12 months (±30 days)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 233
percentage of participants | 0.4 [0.0 to 2.4]

41. Secondary Outcome: Index Limb Amputations
Description: as for outcome 39
Time Frame: 24 months (±30 days)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 207
percentage of participants | 1.0 [0.1 to 3.4]

42. Secondary Outcome: Index Limb Amputations
Description: as for outcome 39
Time Frame: 36 months (±30 days)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 173
percentage of participants | 1.2 [0.1 to 4.1]

43. Secondary Outcome: Quality of Life Assessed (QoL) by SF-12 Questionnaire
Description: The Medical Outcomes Study 12-Item Short form survey (SF-12) was used to assess generic QoL. SF-12 Health Survey is validated measure using 12 questions to measure functional health and well-being from the patient's point of view. Scores on the scale are 0% (indicating poor perceived health status) to 100% (indicating excellent perceived health status) possible. Physical and mental summary scores from the SF-12 are scaled to a U.S. population mean of 50 and standard deviation of 10 (higher scores are better). Multiple groups have suggested minimum clinically important changes in SF-12 summary scores to be greater than 2-2.5 points, and moderate changes to be greater than 5 points.
Time Frame: Baseline
Population: Per ITT set.
  Patients are included in the QoL endpoint if:
  They completed the SF-12 Questionnaire prior to the study procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 264
units on a scale
  Physical Summary Scale | 31.83 (10.11)
  Mental Summary Scale | 49.25 (11.86)

44. Secondary Outcome: Quality of Life Assessed by SF-12 Questionnaire
Description: The Medical Outcomes Study 12-Item Short form survey (SF-12) was used to assess generic QoL.SF-12 Health Survey is validated measure using 12 questions to measure functional health and well-being from the patient's point of view. Scores on the scale are 0% (indicating poor perceived health status) to 100% (indicating excellent perceived health status) possible. Physical and mental summary scores from the SF-12 are scaled to a U.S. population mean of 50 and standard deviation of 10 (higher scores are better). Multiple groups have suggested minimum clinically important changes in SF-12 summary scores to be greater than 2-2.5 points, and moderate changes to be greater than 5 points.
Time Frame: 6 Months (± 14 Days)
Population: Per ITT set.
  Patients are included in the QoL endpoint if:
  They completed the follow-up visit and the SF-12 Questionnaire at the visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 233
units on a scale
  Physical Summary Scale | 38.90 (11.59)
  Mental Summary Scale | 51.51 (11.06)

45. Secondary Outcome: Quality of Life Assessed by SF-12 Questionnaire
Description: as for outcome 44
Time Frame: 12 Months (± 30 Days)
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 229
units on a scale
  Physical Summary Scale | 39.62 (11.03)
  Mental Summary Scale | 51.20 (10.37)

46. Secondary Outcome: Quality of Life Assessed by Peripheral Artery Questionnaire (PAQ): Physical Limitation
Description: The PAQ assesses Peripheral arterial disease (PAD)-related physical limitation, symptoms, quality of life, social function and treatment satisfaction on 0-100 scales; higher scores are better. A threshold of 8 points has been proposed as a minimum clinically important difference for the PAQ summary scale.
Time Frame: Baseline
Population: Per ITT set.
  Patients are included in the QoL endpoint if:
  They completed the PAQ Questionnaire prior to the study procedure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 256
units on a scale | 26.16 (23.06)

47. Secondary Outcome: Quality of Life Assessed by Peripheral Artery Questionnaire (PAQ): Physical Limitation
Description: The PAQ assesses PAD-related physical limitation, symptoms, quality of life, social function and treatment satisfaction on 0-100 scales; higher scores are better. A threshold of 8 points has been proposed as a minimum clinically important difference for the PAQ summary scale.
Time Frame: 6 months (± 14 Days)
Population: Per ITT set.
  Patients are included in the QoL endpoint if:
  They completed the follow-up visit and the PAQ Questionnaire at the visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 209
units on a scale | 52.85 (31.72)

48. Secondary Outcome: Quality of Life Assessed by Peripheral Artery Questionnaire (PAQ): Physical Limitation
Description: as for outcome 47
Time Frame: 12 months (± 30 Days)
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 206
units on a scale | 56.47 (28.82)

49. Secondary Outcome: Quality of Life Assessed by Peripheral Artery Questionnaire (PAQ): Symptoms
Description: as for outcome 47
Time Frame: Baseline
Population: as for outcome 46
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 264
units on a scale | 37.10 (24.40)

50. Secondary Outcome: Quality of Life Assessed by Peripheral Artery Questionnaire (PAQ): Symptoms
Description: as for outcome 47
Time Frame: 6 months (± 14 Days)
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 231
units on a scale | 69.99 (29.25)

51. Secondary Outcome: Quality of Life Assessed by Peripheral Artery Questionnaire (PAQ): Symptoms
Description: as for outcome 47
Time Frame: 12 months (± 30 Days)
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 230
units on a scale | 72.00 (27.71)

52. Secondary Outcome: Quality of Life Assessed by Peripheral Artery Questionnaire (PAQ): Symptom Stability
Description: as for outcome 47
Time Frame: Baseline
Population: as for outcome 46
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 264
units on a scale | 39.02 (21.53)

53. Secondary Outcome: Quality of Life Assessed by Peripheral Artery Questionnaire (PAQ): Symptom Stability
Description: as for outcome 47
Time Frame: 6 months (± 14 Days)
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 232
units on a scale | 55.17 (23.38)

54. Secondary Outcome: Quality of Life Assessed by Peripheral Artery Questionnaire (PAQ): Symptom Stability
Description: as for outcome 47
Time Frame: 12 months (± 30 Days)
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 229
units on a scale | 52.62 (20.65)

55. Secondary Outcome: Quality of Life Assessed by Peripheral Artery Questionnaire (PAQ): Social Limitation
Description: as for outcome 47
Time Frame: Baseline
Population: as for outcome 46
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 261
units on a scale | 48.02 (28.13)

56. Secondary Outcome: Quality of Life Assessed by Peripheral Artery Questionnaire (PAQ): Social Limitation
Description: as for outcome 47
Time Frame: 6 months (± 14 Days)
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 211
units on a scale | 73.16 (29.30)

57. Secondary Outcome: Quality of Life Assessed by Peripheral Artery Questionnaire (PAQ): Social Limitation
Description: as for outcome 47
Time Frame: 12 months (± 30 Days)
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 211
units on a scale | 76.01 (25.60)

58. Secondary Outcome: Quality of Life Assessed by Peripheral Artery Questionnaire (PAQ): Treatment Satisfaction
Description: as for outcome 47
Time Frame: Baseline
Population: as for outcome 46
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 264
units on a scale | 86.46 (18.77)

59. Secondary Outcome: Quality of Life Assessed by Peripheral Artery Questionnaire (PAQ): Treatment Satisfaction
Description: as for outcome 47
Time Frame: 6 months (± 14 Days)
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 232
units on a scale | 87.41 (19.22)

60. Secondary Outcome: Quality of Life Assessed by Peripheral Artery Questionnaire (PAQ): Treatment Satisfaction
Description: as for outcome 47
Time Frame: 12 months (± 30 Days)
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 230
units on a scale | 88.48 (18.07)

61. Secondary Outcome: Quality of Life Assessed by Peripheral Artery Questionnaire (PAQ): Quality of Life
Description: as for outcome 47
Time Frame: Baseline
Population: as for outcome 46
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 264
units on a scale | 35.23 (23.87)

62. Secondary Outcome: Quality of Life Assessed by Peripheral Artery Questionnaire (PAQ): Quality of Life
Description: as for outcome 47
Time Frame: 6 months (± 14 Days)
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 232
units on a scale | 68.70 (29.15)

63. Secondary Outcome: Quality of Life Assessed by Peripheral Artery Questionnaire (PAQ): Quality of Life
Description: as for outcome 47
Time Frame: 12 months (± 30 Days)
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 230
units on a scale | 70.27 (27.00)

64. Secondary Outcome: Quality of Life Assessed by Peripheral Artery Questionnaire (PAQ): Summary Score
Description: as for outcome 47
Time Frame: Baseline
Population: as for outcome 46
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 264
units on a scale | 36.91 (20.94)

65. Secondary Outcome: Quality of Life Assessed by Peripheral Artery Questionnaire (PAQ): Summary Score
Description: as for outcome 47
Time Frame: 6 months (± 14 Days)
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 232
units on a scale | 66.89 (25.95)

66. Secondary Outcome: Quality of Life Assessed by Peripheral Artery Questionnaire (PAQ): Summary Score
Description: as for outcome 47
Time Frame: 12 months (± 30 Days)
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 230
units on a scale | 69.09 (23.19)

67. Secondary Outcome: Clinical Category: Rutherford Becker
Description: Category and Clinical Description
  0 = Asymptomatic, no hemodynamically significant occlusive disease, 1 = Mild claudication, 2 = Moderate claudication, 3 = Severe claudication, 4 = Ischemic rest pain, 5 = Minor tissue loss, non-healing ulcer, or focal gangrene with diffuse pedal ischemia, 6 = Major tissue loss, extending above transmetatarsal level, functional foot no longer salvageable.
  Claudication is defined as a pain, cramps, fatigue, or equivalent in leg muscles occurring during walking that results from inadequate blood supply, usually due to atherosclerotic arterial obstruction.
Time Frame: Baseline
Population: Per ITT Set. Patients are included in the Rutherford Becker Score if the Rutherford Becker Classification was performed prior to the Study procedure.
Measure: Number; unit: percentage of limbs
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 264
percentage of limbs
  Asymptomatic | 0
  Mild Claudication | 0
  Moderate Claudication | 37.5
  Severe Claudication | 57.2
  Ischemic Rest Pain | 5.3
  Minor Tissue Loss | 0
  Major Tissue Loss | 0

68. Secondary Outcome: Clinical Category: Rutherford Becker
Description: as for outcome 67
Time Frame: 1 Month (± 7 Days)
Population: Per ITT Set. Patients are included in the Rutherford Becker Score if they completed their visit and Rutherford Becker Classification was performed
Measure: Number; unit: percentage of limbs
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 259
percentage of limbs
  Asymptomatic | 69.9
  Mild Claudication | 23.9
  Moderate Claudication | 5.0
  Severe Claudication | 1.2
  Ischemic Rest Pain | 0
  Minor Tissue Loss | 0
  Major Tissue Loss | 0

69. Secondary Outcome: Clinical Category: Rutherford Becker
Description: as for outcome 67
Time Frame: 12 Months (± 30 Days)
Population: as for outcome 68
Measure: Number; unit: percentage of limbs
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 230
percentage of limbs
  Asymptomatic | 64.3
  Mild Claudication | 18.7
  Moderate Claudication | 13.9
  Severe Claudication | 2.2
  Ischemic Rest Pain | 0
  Minor Tissue Loss | 0.9
  Major Tissue Loss | 0

70. Secondary Outcome: Clinical Category: Rutherford Becker
Description: as for outcome 67
Time Frame: 24 Months (± 30 Days)
Population: as for outcome 68
Measure: Number; unit: percentage of limbs
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 203
percentage of limbs
  Asymptomatic | 68.0
  Mild Claudication | 17.7
  Moderate Claudication | 10.3
  Severe Claudication | 2.0
  Ischemic Rest Pain | 0
  Minor Tissue Loss | 2.0
  Major Tissue Loss | 0

71. Secondary Outcome: Clinical Category: Rutherford Becker
Description: as for outcome 67
Time Frame: 36 Months (± 30 Days)
Population: as for outcome 68
Measure: Number; unit: percentage of limbs
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 169
percentage of limbs
  Asymptomatic | 72.2
  Mild Claudication | 16.0
  Moderate Claudication | 8.3
  Severe Claudication | 2.4
  Ischemic Rest Pain | 0
  Minor Tissue Loss | 1.2
  Major Tissue Loss | 0

72. Secondary Outcome: Clinical Improvement Compared With Baseline: Rutherford Becker Scale
Description: Clinical Improvement Compared With Baseline
  Grade +3 = Markedly Improved, Grade +2 = Moderately Improved, Grade +1 = Minimally Improved, Grade 0 = No Change, Grade -1 = Mildly Worse, Grade -2 = Moderately Worsening, Grade -3 = Markedly Worsening
Time Frame: 1 month (± 7 Days)
Population: Per ITT Set. Patients are included in the Rutherford Becker Score if :They had a baseline Rutherford Becker Classification performed prior to the study procedure.They completed their visit and Rutherford Becker Classification was performed.
Measure: Number; unit: percentage of limbs
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 259
percentage of limbs
  Grade +3 Markedly Improved | 68.0
  Grade +2 Moderately Improved | 23.2
  Grade +1 Minimally Improved | 6.2
  Grade 0 No Change | 2.7
  Grade -1 Mildly Worse | 0
  Grade -2 Moderately Worsening | 0
  Grade -3 Markedly Worsening | 0

73. Secondary Outcome: Clinical Improvement Compared With Baseline: Rutherford Becker Scale
Description: as for outcome 72
Time Frame: 12 Months (± 30 Days)
Population: as for outcome 72
Measure: Number; unit: percentage of limbs
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 230
percentage of limbs
  Grade +3 Markedly Improved | 53.5
  Grade +2 Moderately Improved | 24.3
  Grade +1 Minimally Improved | 11.3
  Grade 0 No Change | 8.3
  Grade -1 Mildly Worse | 1.3
  Grade -2 Moderately Worsening | 0.9
  Grade -3 Markedly Worsening | 0.4

74. Secondary Outcome: Clinical Improvement Compared With Baseline: Rutherford Becker Scale
Description: as for outcome 72
Time Frame: 24 Months (± 30 Days)
Population: as for outcome 72
Measure: Number; unit: percentage of limbs
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 203
percentage of limbs
  Grade +3 Markedly Improved | 56.7
  Grade +2 Moderately Improved | 25.1
  Grade +1 Minimally Improved | 7.4
  Grade 0 No Change | 4.4
  Grade -1 Mildly Worse | 1.5
  Grade -2 Moderately Worsening | 3.4
  Grade -3 Markedly Worsening | 1.5

75. Secondary Outcome: Clinical Improvement Compared With Baseline: Rutherford Becker Scale
Description: as for outcome 72
Time Frame: 36 Months (± 30 Days)
Population: as for outcome 72
Measure: Number; unit: percentage of limbs
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 167
percentage of limbs
  Grade +3 Markedly Improved | 65.9
  Grade +2 Moderately Improved | 19.8
  Grade +1 Minimally Improved | 6.6
  Grade 0 No Change | 6.0
  Grade -1 Mildly Worse | 0.6
  Grade -2 Moderately Worsening | 0.0
  Grade -3 Markedly Worsening | 1.2

76. Secondary Outcome: Exercise Tolerance Test: Claudication Pain Distance
Description: Absolute Claudication Distance (ACD) for this study was determined by the point of termination or maximum distance walked on the treadmill due to claudication.
Time Frame: Baseline
Population: Per ITT set. The denominator for exercise testing considers factors such as: patient flow to the physician performing the procedure making it difficult to get a baseline treadmill test; patients with bilateral, multilevel peripheral disease and other underlying diseases and other factors such as age could impact their ability to exercise.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 21
meters | 82.32 (62.09)

77. Secondary Outcome: Exercise Tolerance Test: Claudication Pain Distance
Description: as for outcome 76
Time Frame: 1 month (± 7 Days)
Population: as for outcome 76
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 17
meters | 158.87 (140.07)

78. Secondary Outcome: Exercise Tolerance Test: Claudication Pain Distance
Description: as for outcome 76
Time Frame: 12 months
Population: as for outcome 76
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 19
meters | 158.53 (134.95)

79. Secondary Outcome: Exercise Tolerance Test: Claudication Pain Time (CPT)
Description: as for outcome 76
Time Frame: Baseline
Population: as for outcome 76
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 23
seconds | 117.59 (88.41)

80. Secondary Outcome: Exercise Tolerance Test: Claudication Pain Time (CPT)
Description: as for outcome 76
Time Frame: 1 month (± 7 Days)
Population: as for outcome 76
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 17
seconds | 188.12 (151.58)

81. Secondary Outcome: Exercise Tolerance Test: Claudication Pain Time (CPT)
Description: as for outcome 76
Time Frame: 12 months (± 30 Days)
Population: as for outcome 76
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 19
seconds | 195.58 (158.57)

82. Secondary Outcome: Exercise Tolerance Test: Maximal Walking Distance
Description: as for outcome 76
Time Frame: Baseline
Population: as for outcome 76
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 23
meters | 195.38 (107.67)

83. Secondary Outcome: Exercise Tolerance Test: Maximal Walking Distance
Description: as for outcome 76
Time Frame: 1 month (± 7 Days)
Population: as for outcome 76
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 18
meters | 294.18 (244.24)

84. Secondary Outcome: Exercise Tolerance Test: Maximal Walking Distance
Description: as for outcome 76
Time Frame: 12 months (± 30 Days)
Population: as for outcome 76
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 19
meters | 262.61 (141.58)

85. Secondary Outcome: Exercise Tolerance Test: Maximal Walking Time
Description: as for outcome 76
Time Frame: Baseline
Population: as for outcome 76
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 23
seconds | 245.71 (136.00)

86. Secondary Outcome: Exercise Tolerance Test: Maximal Walking Time
Description: as for outcome 76
Time Frame: 1 month (± 7 Days)
Population: as for outcome 76
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 18
seconds | 345.22 (255.76)

87. Secondary Outcome: Exercise Tolerance Test: Maximal Walking Time
Description: as for outcome 76
Time Frame: 12 months (± 30 Days)
Population: as for outcome 76
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Supera® Peripheral Stent System
Number analyzed (Participants) | 19
seconds | 317.53 (159.38)

ADVERSE EVENTS:
Time Frame: 3 Years
Groups:
- Supera® Peripheral Stent System ITT: Implantation of Supera stent using the Supera® Peripheral Stent System.
  ITT population consisted of 264 subjects.
- Supera® Peripheral Stent System Roll-in: Implantation of Supera stent using the Supera® Peripheral Stent System.
  There were a total of 61 roll-in subjects.
Arm/Group | Supera® Peripheral Stent System ITT | Supera® Peripheral Stent System Roll-in
Serious Adverse Events (participants affected / at risk) | 151/264 | 36/61
Other Adverse Events (participants affected / at risk) | 211/264 | 51/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supera® Peripheral Stent System ITT (N=264) | Supera® Peripheral Stent System Roll-in (N=61)
Anaemia (Blood and lymphatic system disorders) | 9 (9) | 2 (2)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 10 (10) | 1 (1)
Angina pectoris (Cardiac disorders) | 3 (4) | 1 (1)
Angina unstable (Cardiac disorders) | 7 (9) | 2 (2)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 4 (4)
Atrial flutter (Cardiac disorders) | 3 (3) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 3 (3) | 0 (0)
Cardiac failure (Cardiac disorders) | 3 (3) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 9 (14) | 2 (4)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 17 (22) | 2 (3)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
In-stent coronary artery restenosis (Cardiac disorders) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 3 (5) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 2 (2) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Spondylolisthesis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 8 (8) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Reflux gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Brain death (General disorders) | 1 (1) | 0 (0)
Cardiac death (General disorders) | 1 (1) | 0 (0)
Catheter site haematoma (General disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 2 (2)
Chest pain (General disorders) | 15 (18) | 3 (3)
Death (General disorders) | 3 (3) | 0 (0)
Multi-organ failure (General disorders) | 2 (2) | 0 (0)
Necrosis (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Iodine allergy (Immune system disorders) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (2)
Diverticulitis (Infections and infestations) | 3 (3) | 0 (0)
Gangrene (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Meningitis viral (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 5 (8) | 2 (2)
Pneumonia (Infections and infestations) | 10 (11) | 2 (2)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1)
Device malfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 17 (24) | 3 (4)
Medical device complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Open wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural swelling (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pubic rami fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Renal injury (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stent occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular graft complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetic foot (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (8) | 2 (3)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 3 (4) | 0 (0)
Cerebellar haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 2 (4)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Facial palsy (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 2 (2) | 0 (0)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 4 (4) | 3 (4)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0)
Mental status changes (Psychiatric disorders) | 3 (3) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (2) | 0 (0)
Malignant renal hypertension (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 3 (3) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 3 (3) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (4)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (5)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Large intestine anastomosis (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Arterial restenosis (Vascular disorders) | 1 (1) | 0 (0)
Arterial stenosis limb (Vascular disorders) | 1 (1) | 1 (1)
Arterial thrombosis limb (Vascular disorders) | 2 (2) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Arteriovenous fistula (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 1 (1)
Femoral arterial stenosis (Vascular disorders) | 4 (4) | 3 (3)
Femoral artery occlusion (Vascular disorders) | 3 (3) | 0 (0)
Haemorrhage (Vascular disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Iliac artery stenosis (Vascular disorders) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 17 (20) | 4 (5)
Leriche syndrome (Vascular disorders) | 1 (1) | 0 (0)
Malignant hypertension (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 11 (14) | 2 (4)
Peripheral artery aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery dissection (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 7 (8) | 2 (2)
Peripheral vascular disorder (Vascular disorders) | 12 (17) | 2 (2)
Vascular pseudoaneurysm (Vascular disorders) | 1 (1) | 0 (0)
Venous stasis (Vascular disorders) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Graft dysfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carotid artery disease (Nervous system disorders) | 1 (1) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supera® Peripheral Stent System ITT (N=264) | Supera® Peripheral Stent System Roll-in (N=61)
Anaemia (Blood and lymphatic system disorders) | 15 (16) | 2 (2)
Coronary artery disease (Cardiac disorders) | 17 (22) | 2 (3)
Catheter site haematoma (General disorders) | 16 (17) | 3 (4)
Chest pain (General disorders) | 20 (25) | 6 (6)
Oedema peripheral (General disorders) | 19 (21) | 7 (8)
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 28 (37) | 6 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 41 (51) | 16 (20)
Femoral artery dissection (Vascular disorders) | 29 (32) | 6 (6)
Intermittent claudication (Vascular disorders) | 39 (52) | 7 (13)
Peripheral arterial occlusive disease (Vascular disorders) | 17 (22) | 3 (5)
Peripheral vascular disorder (Vascular disorders) | 16 (24) | 3 (4)
Atrial fibrillation (Cardiac disorders) | 4 (5) | 4 (5)
Cardiac failure congestive (Cardiac disorders) | 10 (15) | 4 (6)
Nausea (Gastrointestinal disorders) | 8 (9) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (13) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (12) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 6 (10)
Hypertension (Vascular disorders) | 7 (7) | 3 (3)
Pneumonia (Infections and infestations) | 10 (11) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less